CLINICAL TRIAL: NCT04601220
Title: Social Media, Smartphone Use and Self-harm in Young People
Acronym: 3S-YP
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 269104
Record Dates: First submitted 2020-10-07; First posted 2020-10-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-10

CONDITIONS: Self-Harm, Deliberate
Keywords: Young adult; Adolescent; Social media; Smartphone; Mental health
MeSH Terms: conditions — Self-Injurious Behavior; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Self-harm is when somebody hurts their body as a way of coping with difficult feelings. Self-harm is becoming increasingly common in young people, particularly in adolescent females. The rise in self-harm has been linked to increasing use of social media and internet technology among young people. However, the evidence is limited to associations with poorer mental health outcomes rather than identifying particular aspects of using these technologies that can negatively impact on mental health.

This study aims to investigate how the use of social media and a smartphone may increase the risk of self-harm in young people by exploring changes in usage in the period leading up to an episode of self-harm. The information from this study will allow us to understand whether there are certain behaviours that are more likely to occur before an episode of self-harm. This will inform new strategies to identify and provide support to vulnerable young people. For example, linking young people with crisis support or empowering young people to make changes, manage their own risks and build resilience.

This study will recruit young people aged 13-25 years old who have accessed mental health services provided by an NHS Trust in South-East London. Young people will be invited to provide information on their mental health and social media and smartphone use over a period of six months.

ELIGIBILITY:
Inclusion criteria

* Identified via SLaM's C4C patient research participation register or referral to the study team by their clinician.
* Aged 13-25 years old at the time of study approach.
* Accessed mental health services at SLaM in the last 12 months.
* Has capacity to consent (and an adult with parental responsibility for young people aged 13-15 years old). Mental capacity will be assumed unless evidence from a clinician or during contact with the study team suggests otherwise.

Exclusion criteria

* Unable to complete the questionnaires via the study software application or online survey platform.
* Admitted to an inpatient psychiatric ward, sectioned under the Mental Health Act or in prison at the time of approach.
* Clinician advises it is not appropriate to approach.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Self-harm event | 6 months
  Self-reported and clinician-reported self-harm events

SECONDARY OUTCOMES:
Sleep disturbance symptoms | 6 months
  Symptoms of sleep disturbance measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form V1.0 4a / Pediatric Sleep Disturbance Short Form V1.0 4a. Scores range between 4-20, with higher scores indicative of possible sleep disturbance.
Depression symptoms | 6 months
  Symptoms of depression measured using the Patient Health Questionnaire. Scores range between 0-27, with higher scores indicative of possible depression.
Anxiety symptoms | 6 months
  Symptoms of anxiety measured using the Generalized Anxiety Disorder Scale. Scores range between 0-21, with higher scores indicative of possible generalised anxiety disorder.
Loneliness symptoms | 6 months
  Symptoms of loneliness measured using the Three-Item Loneliness Scale. Scores range between 3-9, with higher scores indicative of possible loneliness.
Experiences of being bullied | 6 months
  Experiences of being bullied measured using an Eight-Item Bullying Checklist derived from the Revised Olweus Bully/Victim Questionnaire. Scores range between 8-40, with higher scores indicative of more experiences of being bullied.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Dutta, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be made available to other researchers.

REFERENCES:
- [Background] Bye A, Carter B, Leightley D, Trevillion K, Liakata M, Branthonne-Foster S, Williamson G, Zenasni Z, Dutta R. Observational prospective study of social media, smartphone use and self-harm in a clinical sample of young people: study protocol. BMJ Open. 2023 Feb 1;13(2):e069748. doi: 10.1136/bmjopen-2022-069748. PMID 36725102
- [Background] Bye A, Carter B, Leightley D, Trevillion K, Liakata M, Branthonne-Foster S, Cross S, Zenasni Z, Carr E, Williamson G, Vega Viyuela A, Dutta R. Cohort profile: The Social media, smartphone use and Self-harm in Young People (3S-YP) study-A prospective, observational cohort study of young people in contact with mental health services. PLoS One. 2024 May 22;19(5):e0299059. doi: 10.1371/journal.pone.0299059. eCollection 2024. PMID 38776261
- [Derived] Bye A, Trevillion K, Wilson-Lemoine E, Leightley D, Carter B, Liakata M, Hopper J, Dutta R. Visual content and thematic analyses of images shared on social media before and after episodes of self-harm in a UK clinical youth sample. BMJ Open. 2026 Jan 19;16(1):e103456. doi: 10.1136/bmjopen-2025-103456. PMID 41554580
- [Derived] Bye A, Wilson-Lemoine E, Trevillion K, Carter B, Dutta R. Factors that affect clinical youth engagement in digital mental health research: a qualitative sub-study nested within a prospective cohort study. BMC Med Res Methodol. 2025 Apr 30;25(1):118. doi: 10.1186/s12874-025-02571-9. PMID 40307751
- See also: Related Info — https://www.3syp.com